CLINICAL TRIAL: NCT05013931
Title: Short-term Effect of COVID-19 Vaccine on Blood Pressure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kelvin KF Tsoi, Associate Professor, Chinese University of Hong Kong
Other Study IDs: 2021.449
Record Dates: First submitted 2021-08-17; First posted 2021-08-19 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Covid19; Blood Pressure
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate short-term effect of COVID-19 vaccination on blood pressure by conducting 24-hour ABPM

DETAILED DESCRIPTION:
Safety of coronavirus disease 19 (COVID-19) vaccines has been a concern. Despite safety profile of different vaccines demonstrated in phase 2/3 trials, there has been evolving evidence on adverse effects of some particular COVID-19 vaccines. One of the mostly known example is vaccine-induced thrombotic thrombocytopenia (VITT). Apart from the thrombotic risk of ChAdOx1 nCoV-19 vaccine, there has been studies providing the preliminary data on effect of mRNA-based COVID-19 vaccine on blood pressure.

A case series report was published on Hypertension in June 2021 on documented stage III hypertension within minutes of vaccination (mRNA vaccines) in a vaccination centre located in Switzerland. The study reported 9 subjects experienced a surge in blood pressure to stage III hypertension after vaccination. Yet the study had a few shortcomings. There was not baseline measurement of blood pressure. Surge of blood pressure shortly after vaccination could be due to nervousness or white coat effect. Thus surge of blood pressure within minutes of vaccination could be not due to vaccination. There was not long-term follow-up on blood pressure measurement after vaccination.

Further to the case series report, another prospective study in Italy investigated effect of mRNA vaccine on blood pressure and heart rate. The study was conducted as a survey. There was 5.3% of respondents (6/113) reported rise of home blood pressure of at least 10mmHg after 1st dose vaccination, compared with home blood pressure prior to vaccination. Among these subjects, 4 of them required anti-hypertensive medication intensification.

Yet there remains lack of evidence and detailed description on effect of COVID-19 vaccines and blood pressure before and after vaccination. Use of ambulatory blood pressure monitoring (ABPM) before and after vaccination helps to understand the details on short-term blood pressure changes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who will be receiving COVID-19 vaccination
* Subjects who understand Chinese to make an informed consent

Exclusion Criteria:

* Skin condition around the cuff not suitable for long term cuff wearing (e.g. severe dermatitis, wound)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants who will be receiving COVID-19 vaccination will be invited to the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
To investigate short-term effect of COVID-19 vaccination on blood pressure by conducting 24-hour ABPM | 1 day